CLINICAL TRIAL: NCT03726775
Title: A Phase II Trial of Radiotherapy (RT)-Durvalumab Without Prophylactic Neck Irradiation in Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Trial Evaluating the Tolerance and Safety of Durvalumab - RT Combination for Treatment in SCCHN
Acronym: REWRITe
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: UNICANCER (Other); Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2018-02
Record Dates: First submitted 2018-10-25; First posted 2018-10-31 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: HNSCC
Keywords: durvalumab; without prophylactic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: IV infusion of durvalumab will start at fixed dose on Day1 of RT and subsequently every 3 weeks during the course of RT. Durvalumab with be continued via IV infusion at a fixed dose for an additional 6 months following RT, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RT-durvalumab (Experimental): durvalumab at fixed dose of 1120 mg on Day1 of RT and every 3 weeks during the RT. Durvalumab with be continued at a fixed dose of 1500 mg every 4 weeks during 6 months following RT.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Infusion of durvalumab during RT and after RT during 6 months
  Other Names: MEDI4736

SUMMARY:
This study evaluate the regional (neck) nodal control of durvalumab in combination with RT restricted to the primary tumor and the immediately adjacent nodal level (i.e. without prophylactic neck irradiation) in N0 patients with SCCHN.

DETAILED DESCRIPTION:
There is a strong rationale for testing this new paradigm of RT for SCCHN without prophylactic neck irradiation, being replaced by immune stimulation via the combination of RT and Programmed Death-1 (PD-L1) inhibition with durvalumab, due to:

* The unmet medical need for new treatments, better tolerated and " as " or " more " effective than the current Standard Of Care (SOC)
* The need to decrease radiation-induced toxicity, especially in fragile patients
* The added toxicity due to elective nodal irradiation
* The strong rationale to combine RT and PD-L1 inhibition
* The potential immune suppressive effect of large field prophylactic neck irradiation

It is hypothesized this innovative concept to be safe in the context of this study for the following reasons:

* The rate of relapse in the neck is expected to be low in Magnetic Resonnance Imaging (MRI) & PET-CT N0 neck
* A non-irradiated neck can be easily monitored, clinically and by imaging
* Most of the potential relapses in the neck are expected to be salvaged by surgery and/or RT
* The preventive irradiation of N0 regions is not anymore performed for others lymphophilic cancers (lymphoma, Non-Small Cell Lung Cancer (NSCLC)).

The combination of durvalumab with RT restricted to the primary tumor site and immediate adjacent nodal area will achieve a similarly regional (nodal) control rate than standard RT including large prophylactic neck irradiation (regional recurrence < 10 %.

This study will include patients with early (T1-T2 N0) or locally advanced SCCHN (T3-4 N0), histologically proven who had not received previous treatment for this setting. The study is designed with the primary objective of demonstrating that RT without large prophylactic irradiation in combination with durvalumab is effective in terms of regional control. All patients will be followed until death or at least 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years with no upper limit
2. Performance Status ECOG 0-2
3. Squamous cell carcinoma, previously untreated
4. T1-T4 with clinical status N0-N1 or N2a-N2b non palpable, with only homolateral lymph node in radiological examinations.
5. Patient with at least one of these fragility criteria :

   o Status ECOG 1 with multiple comorbidities, at least 2 pathologies with grade ≥ 2 (renal and/or cardiac and/or vascular and/or hepatic, and/or,neurologic, and/or pulmonary)

   o Status ECOG = 2

   o Age ≥ 70 , judged unfit with oncogeratric evaluation by EGE (ELAN Geriatric Evaluation) test or unable to receive cisplatine or Carboplatine- 5FU (at least one criteria listed below*)

   * Criteria for determining if a patient is unfit for receiving cisplatine or carbo-5FU :

   - Calculated creatinine clearance ≤ 60 mL/min as determined by the modified. method of Cockcroft and Gault or glomerular filtration rate ≤ 60 mL/min/1.73m² (CKD-EPI method recommended)

   - Haemoglobin < 10 g/dL, aspartate (AST) and alanine transaminase (ALT) more than 2 times the upper limit of the normal range (ULN), serum albumin ≤35 g/L, Absolute neutrophil count ≤ 1 500/μL, platelets ≤ 100 000/μL or total bilirubin ≥ 1.5 mg/dL
   * Cardiac function not compatible with hyperhydration or significant heart disease
   * Weight loss > 15% in 2 months
6. Oral cavity, oropharynx, hypopharynx or larynx
7. Availability of pre-treatment tumor tissue sample (for PD-L1 expression, TILs and immune landscape)
8. Documentation of p16 disease (HPV status for oropharyngeal tumor)
9. Recording of alcohol consumption and smoking history
10. Glomerular filtration rate (GFR) >40 mL/min/1.73m2 (CKD-EPI method recommended) or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula
11. Patient willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations during the follow up period
12. Patient able to understand French and complete the quality of life questionnaires or who can be helped by a support person if necessary.
13. Must have a life expectancy of at least 12 weeks
14. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

1) Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and folliclestimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

2) Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

15. Written informed consent obtained prior to performing any protocol-related procedures, including screening evaluations

Exclusion Criteria:

1. Nasopharyngeal, paranasal sinuses, nasal cavity tumors or thyroid cancers
2. Metastatic disease
3. Active CNS disease
4. Any prior or current treatment for invasive head and neck cancer
5. Any unresolved toxicity NCI CTCAE v5.0 Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the investigator
6. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable
7. History of leptomeningeal carcinomatosis
8. Body weight ≤ 30 kg and/or weight loss of ≥ 15% during the last 4 weeks (except if renutrition with a feeding tube is planned before the onset of treatment or is ongoing)
9. Concurrent treatment with any other systemic anti-cancer therapy that is not specified in the protocol
10. Concomitant treatment with any drug on the prohibited medication list such as live vaccines within 30 days prior to the first dose of IP
11. Known allergy or hypersensitivity reaction to study drug or any of the study drug excipients
12. Prior organ transplantation including allogenic stem-cell transplantation
13. Other severe acute or chronic medical conditions including pneumonitis, pulmonary fibrosis
14. Active autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc])
15. Uncontrolled intercurrent illness, including but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
16. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥ 5 years
    2. Adequately treated non-melanoma skin cancer
    3. Adequately treated carcinoma in situ without evidence of disease
17. History of active primary immunodeficiency
18. Ongoing or active infection including tuberculosis, hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections
    2. Systemic corticosteroids < 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
21. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment
22. Individual deprived of liberty, or under any kind of guardianship
23. Inclusion in another study research on drug or medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Regional (neck) nodal control rate | 1 year
  Cervical Node Control in the non-irradiated N0 neck

SECONDARY OUTCOMES:
Recurrence and control rates analysis | 3, 6, 12, 18, 24 and 36 months
  Estimation of local, regional, locoregional control
Survival analyses | 3, 7, 11, 15, 19, 23, 27, 31, and 36 months post RT
  Estimation of the survival rates and the 95% confidence intervals (95% CI)
Objective Response Rate | 3, 12, 24 et 36 months post RT
  complete or partial response according to RECIST 1.1 criteria
Quality of life QLQC30 | baseline, 3-month, 12-month and 24-month post RT
  To evaluate the effectiveness of support
Quality of life QLQ-H&N35 | baseline, 3-month, 12-month and 24-month post RT
  To evaluate the effectiveness of support

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Sainte Catherine, Avignon
  - Centre Eugene Marquis, Rennes

IPD SHARING:
Plan to Share IPD: Undecided